CLINICAL TRIAL: NCT02601014
Title: Biomarker-Driven Phase-2 Study of Combined Immune Checkpoint Blockade for AR-V7-Expressing Metastatic Castration-Resistant Prostate Cancer (STARVE-PC)
Brief Title: Biomarker-Driven Therapy With Nivolumab and Ipilimumab in Treating Patients With Metastatic Hormone-Resistant Prostate Cancer Expressing AR-V7
Acronym: STARVE-PC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J15119; NCI-2015-01325 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); J15119 (Other: Johns Hopkins University/Sidney Kimmel Cancer Center); IRB00070748 (Other: JHM IRB)
Record Dates: First submitted 2015-08-21; First posted 2015-11-10 (Estimated); Results first posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Prostate Cancer; Recurrent Prostate Carcinoma; Stage IV Prostate Adenocarcinoma
Keywords: Hormone-Resistant Prostate Cancer; Prostate Carcinoma Metastatic in the Bone
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ipilimumab; CTLA-4 Antigen; Nivolumab; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nivolumab and ipilimumab (Experimental): Patients receive nivolumab IV over 60 minutes and ipilimumab IV over 90 minutes every 3 weeks for 12 weeks. Patients then receive nivolumab IV over 60 minutes every 2 weeks for 36 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Biological: Nivolumab
- Enzalutamide plus Nivolumab and Ipilimumab (Experimental): Patients will continue on standard of care enzalutamide, with the addition of nivolumab IV over 60 minutes and ipilimumab IV over 90 minutes every 3 weeks for 12 weeks. Patients then receive nivolumab IV over 60 minutes every 2 weeks for 36 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Biological: Nivolumab; Drug: Enzalutamide

INTERVENTIONS:
Biological: Ipilimumab — Given 1 mg/kg IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy
Biological: Nivolumab — Given 3 mg/kg IV
  Other Names: BMS-936558; MDX-1106; ONO-4538; Opdivo
Drug: Enzalutamide — given orally per standard of care
  Other Names: Xtandi
  Arms: Enzalutamide plus Nivolumab and Ipilimumab

SUMMARY:
This phase II trial studies how well nivolumab and ipilimumab work in treating patients with hormone-resistant prostate cancer that has spread to other places in the body and express androgen receptor-variant-7 (AR-V7). Tumor cells expressing AR-V7 has been shown to be resistant to hormone therapy and some chemotherapy in patients with prostate cancer. Biomarker-driven therapy, such as nivolumab and ipilimumab, may work by blocking key biomarkers or proteins that help tumor cells to escape the immune system surveillance and this may help the immune system to kill tumor cells that express AR-V7.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate
* Metastatic disease as defined by two or more bone metastases confirmed by bone scintigraphy or radiographic soft tissue metastasis
* Detectable circulating tumor cells (CTCs) with detectable AR-V7 splice-variant by reverse transcriptase (RT)-polymerase chain reaction (PCR)

For second cohort (amendment 1):

The most recent therapy must be enzalutamide and enzalutamide will be continued for study duration despite progressive disease. The minimum required dose of Enzalutamide at enrolment should be no less than 80 mg once daily.

* Known castration-resistant disease, defined according to Prostate Cancer Working Group 2 (PCWG2) criteria as:

  * Castrate serum testosterone level: =< 50 ng/dL (=< 1.7 nmol/L)
  * Subjects who have failed initial hormonal therapy, either by orchiectomy or by using a gonadotropin-releasing hormone (GnRH) agonist in combination with an anti-androgen, must first progress through antiandrogen withdrawal prior to being eligible; the minimum timeframe to document failure of anti-androgen withdrawal will be four weeks
  * Serum PSA progression defined as two consecutive increases in PSA over a previous reference value within 6 months of first study treatment, each measurement at least one week apart; serum PSA at screening >= 2 ng/mL OR

    * Documented bone lesions by the appearance of two or more new lesions by bone scintigraphy OR
    * Bidimensionally-measureable soft tissue metastatic lesion assessed by computed tomography (CT) or magnetic resonance imaging (MRI)
* Karnofsky performance status (KPS): >= 70% within 14 days before start of study treatment (Eastern Cooperative Oncology Group [ECOG] =< 1)
* Life expectancy: at least 6 months
* White blood count (WBC) >= 2000/uL
* Neutrophils >= 1500/uL
* Platelets >= 100 x10^3/uL
* Hemoglobin > 9.0 g/dL
* Serum creatinine =< 1.5 x upper limit of normal (ULN) or creatinine clearance (CrCl) >= 40 mL/min (if using the Cockcroft-Gault formula)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 3 x ULN
* Total bilirubin =< 1.5 x ULN (except subjects with Gilbert syndrome, who can have total bilirubin < 3.0 mg/dL)
* Men who are sexually active with women of childbearing potential (WOCBP) must use any contraceptive method with a failure rate of less than 1% per year; men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product
* WOCBP is defined as any female who has experienced menarche and has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal; menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes; in addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/mL
* No evidence (within 5 years) of prior malignancies (except successfully treated basal cell or squamous cell carcinoma of the skin)
* The subject is willing and able to comply with the protocol, and agrees to return to the hospital for follow-up visits and examination
* The subject has been fully informed about the study and has signed the informed consent form and, where appropriate, Health Insurance Portability and Accountability Act (HIPAA) authorization for release of personal health information

  * NOTE: HIPAA authorization may be included in the informed consent or obtained separately

Exclusion Criteria:

* Has received an investigational therapeutic drug within the last 4 weeks prior to start of study treatment, or is scheduled to receive one during the treatment period
* Has received external radiotherapy within the last 4 weeks prior to start of study treatment
* Previous therapy with antiandrogens within 4 weeks
* Patients should be excluded if they have had prior systemic treatment with an anti-programmed cell death protein 1 (PD-1), anti-PD-L1, anti-programmed cell death 1 ligand 2 (PD-L2), anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways
* Symptomatic metastatic disease with signs of rapid progression per investigator's clinical judgment
* Concurrent use of other anticancer agents or treatments, with the following exceptions:

  * Ongoing treatment with luteinizing hormone-releasing hormone (LHRH) agonists or antagonists, denosumab (Prolia) or bisphosphonate (eg, zoledronic acid) is allowed; ongoing treatment should be kept at a stable schedule; however, if medically required, a change of dose, compound, or both is allowed
* Any treatment modalities involving major surgery within 4 weeks prior to the start of study treatment
* Symptomatic nodal disease, i.e. scrotal, penile or leg edema (>= Common Terminology Criteria for Adverse Events [CTCAE] grade 3)
* Patients are excluded if they have active brain metastases or leptomeningeal metastases; subjects with brain metastases are eligible if metastases have been treated and there is no magnetic resonance imaging (MRI) evidence of progression for at least 4 weeks after treatment is complete and within 28 days prior to the first dose of nivolumab administration; there must also be no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration
* Patients should be excluded if they have an active, known or suspected autoimmune disease (e.g. inflammatory bowel disease, rheumatoid arthritis, autoimmune hepatitis, lupus, celiac disease); subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration; inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
* Permitted therapies include topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption); physiologic replacement doses of systemic corticosteroids are permitted, even if > 10 mg/day prednisone equivalents; a brief course of corticosteroids for prophylaxis (eg, contrast dye allergy) or for treatment of nonautoimmune conditions (e.g. delayed-type hypersensitivity reaction caused by contact allergen) is permitted
* Drugs with a predisposition to hepatoxicity should be used with caution in patients treated with nivolumab-containing regimen
* Patients should be excluded if they have a positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection
* Patients should be excluded if they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Allergies and adverse drug reaction
* History of allergy to study drug components
* History of severe hypersensitivity reaction to any monoclonal antibody
* Other primary tumor (other than castration-resistant prostate cancer [CRPC]) including hematological malignancy present within the last 5 years (except non-melanoma skin cancer or low-grade superficial bladder cancer)
* Has imminent or established spinal cord compression based on clinical findings and/or MRI
* Any other serious illness or medical condition that would, in the opinion of the investigator, make this protocol unreasonably hazardous, including, but not limited to:

  * Any uncontrolled infection
  * Cardiac failure NYHA (New York Heart Association) III or IV
  * Crohn's disease or ulcerative colitis
  * Bone marrow dysplasia
  * Known allergy to any of the compounds under investigation
  * Unmanageable fecal incontinence

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2021-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Antonarakis, Principal Investigator — Johns Hopkins University/Sidney Kimmel Cancer Center
Locations (1):
- Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Boudadi K, Suzman DL, Anagnostou V, Fu W, Luber B, Wang H, Niknafs N, White JR, Silberstein JL, Sullivan R, Dowling D, Harb R, Nirschl TR, Veeneman BA, Tomlins SA, Wang Y, Jendrisak A, Graf RP, Dittamore R, Carducci MA, Eisenberger MA, Haffner MC, Meeker AK, Eshleman JR, Luo J, Velculescu VE, Drake CG, Antonarakis ES. Ipilimumab plus nivolumab and DNA-repair defects in AR-V7-expressing metastatic prostate cancer. Oncotarget. 2018 Jun 19;9(47):28561-28571. doi: 10.18632/oncotarget.25564. eCollection 2018 Jun 19. PMID 29983880
- [Result] Shenderov E, Boudadi K, Fu W, Wang H, Sullivan R, Jordan A, Dowling D, Harb R, Schonhoft J, Jendrisak A, Carducci MA, Eisenberger MA, Eshleman JR, Luo J, Drake CG, Pardoll DM, Antonarakis ES. Nivolumab plus ipilimumab, with or without enzalutamide, in AR-V7-expressing metastatic castration-resistant prostate cancer: A phase-2 nonrandomized clinical trial. Prostate. 2021 May;81(6):326-338. doi: 10.1002/pros.24110. Epub 2021 Feb 26. PMID 33636027

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two subjects were screen failures.
Period: Overall Study
Arm/Group | Nivolumab and Ipilimumab | Enzalutamide Plus Nivolumab and Ipilimumab
Started | 15 | 15
Completed | 5 | 3
Not Completed | 10 | 12
Not completed — Adverse Event | 3 | 3
Not completed — Death | 3 | 1
Not completed — Disease progression | 4 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab and Ipilimumab | Enzalutamide Plus Nivolumab and Ipilimumab | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 3 | 10
  >=65 years | 8 | 12 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 15 | 15 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white | 14 | 13 | 27
  non-white | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Change in PSA Response
Description: Number of participants with greater than 50% decline in PSA from start of treatment, sustained for >= 4 weeks, as defined by Prostate Cancer Working Group 2 (PCWG2) criteria.
Time Frame: up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab and Ipilimumab | Enzalutamide Plus Nivolumab and Ipilimumab
Number analyzed (Participants) | 15 | 15
Participants | 2 | 0

2. Secondary Outcome: Durable Progression Free Survival (PFS)
Description: Number of participants with PFS >= 24 weeks. PFS is described as number of weeks from start of treatment until first evidence of clinical radiographic progression, or death.
Time Frame: up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab and Ipilimumab | Enzalutamide Plus Nivolumab and Ipilimumab
Number analyzed (Participants) | 15 | 15
Participants | 3 | 4

3. Secondary Outcome: Number of Participants Experiencing Adverse Events
Description: Number of participants experiencing Grade 3-4 adverse events, Grade 3-4 immune-related AEs (irAEs), as defined by National Cancer Institute (NIH) CTCAE version 4.0
Time Frame: up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab and Ipilimumab | Enzalutamide Plus Nivolumab and Ipilimumab
Number analyzed (Participants) | 15 | 15
Participants
  Grade 3-4 | 7 | 8
  Grade 3-4 irAE | 5 | 7
  Grade 3-4 AE leading to treatment discontinuation | 6 | 3

4. Secondary Outcome: Objective Response Rate (ORR)
Description: Number of participants with complete response (CR) or partial response (PR) in measurable soft tissue lesions, as defined by RECIST version 1.1
Time Frame: up to 3 years
Population: Only 8/15 in Arm 1 and 9/15 in Arm 2 were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab and Ipilimumab | Enzalutamide Plus Nivolumab and Ipilimumab
Number analyzed (Participants) | 8 | 9
Participants | 2 | 0

5. Secondary Outcome: Overall Survival
Description: Number of months alive after start of treatment.
Time Frame: up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab and Ipilimumab | Enzalutamide Plus Nivolumab and Ipilimumab
Number analyzed (Participants) | 15 | 15
months | 8.2 [5.5 to 10.4] | 14.2 [8.5 to NA] — Insufficient number of participants with events.

6. Secondary Outcome: Progression Free Survival (PFS)
Description: Number of months from start of treatment until first evidence of progression, as defined by based on RECIST version 1.1 and PCWG2
Time Frame: up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab and Ipilimumab | Enzalutamide Plus Nivolumab and Ipilimumab
Number analyzed (Participants) | 15 | 15
months | 3.7 [2.8 to 7.5] | 2.9 [1.3 to 5.8]

7. Secondary Outcome: Number of Participants With Change in AR-V7 Expression
Description: Change in AR-V7 expression is defined as converting from AR-V7-positive to AR-V7-negative during treatment.
Time Frame: up to 3 years
Population: Data was not collected for this outcome measure.
Arm/Group | Nivolumab and Ipilimumab | Enzalutamide Plus Nivolumab and Ipilimumab
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: PSA-PFS
Description: Number of months until >= 25% or >=2 ng/mL increase in PSA, as defined per PCWG2 criteria
Time Frame: up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab and Ipilimumab | Enzalutamide Plus Nivolumab and Ipilimumab
Number analyzed (Participants) | 15 | 15
months | 3.0 [2.1 to NA] — Insufficient number of participants with events. | 2.7 [2.1 to 5.9]

9. Secondary Outcome: Response Duration in Patients With Objective Response
Description: Number of months from first evidence of response until progression.
Time Frame: up to 12 months
Population: Data was not evaluable for this outcome measure.
Arm/Group | Nivolumab and Ipilimumab | Enzalutamide Plus Nivolumab and Ipilimumab
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Number of Participants With Change in AR-V7 Expression as Expressed by AR-V7 to Full Length AR Ratio Converting From AR-V7-positive to -Negative With Changes in AR-V7 Expression
Description: Change in AR-V7 is described as converting from AR-V7-positive to -negative, expressed as a ratio of AR-V7 to full-length AR (AR-FL)
Time Frame: up to 3 years
Population: Data was not collected for this outcome measure.
Arm/Group | Nivolumab and Ipilimumab | Enzalutamide Plus Nivolumab and Ipilimumab
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 3 years
Arm/Group | Nivolumab and Ipilimumab | Enzalutamide Plus Nivolumab and Ipilimumab
All-Cause Mortality (participants affected / at risk) | 9/15 | 2/15
Serious Adverse Events (participants affected / at risk) | 6/15 | 5/15
Other Adverse Events (participants affected / at risk) | 15/15 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab and Ipilimumab (N=15) | Enzalutamide Plus Nivolumab and Ipilimumab (N=15)
intracranial hemorrhage (Nervous system disorders) | 2 (2) | 0 (0)
chronic subdural hematoma (Vascular disorders) | 1 (1) | 0 (0)
elevated bilirubin (Investigations) | 1 (1) | 0 (0)
hepatitis (Infections and infestations) | 1 (1) | 0 (0)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
elevated liver function test (Hepatobiliary disorders) | 1 (1) | 0 (0)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
allergic reaction to amoxicillin (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
generalized weakness (General disorders) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
infusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
fever (General disorders) | 0 (0) | 1 (1)
lactate elevation (Investigations) | 0 (0) | 1 (1)
expressive aphasia (Psychiatric disorders) | 0 (0) | 1 (1)
dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
eosinophilia (Investigations) | 0 (0) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Addison's disease (Endocrine disorders) | 0 (0) | 1 (1)
hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (1)
immune related colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypophysitis (Endocrine disorders) | 0 (0) | 1 (1)
central adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab and Ipilimumab (N=15) | Enzalutamide Plus Nivolumab and Ipilimumab (N=15)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (16) | 6 (12)
edema (General disorders) | 4 (5) | 1 (1)
anemia (Blood and lymphatic system disorders) | 8 (14) | 5 (7)
Alkaline phosphatase increased (Hepatobiliary disorders) | 3 (5) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 1 (1)
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
leg weakness (General disorders) | 2 (2) | 0 (0)
difficulty urinating (Renal and urinary disorders) | 2 (2) | 2 (2)
Alanine Aminotransferase increased (Investigations) | 3 (6) | 3 (3)
lipase increased (Investigations) | 4 (4) | 2 (6)
hematocrit count decreased (Blood and lymphatic system disorders) | 7 (8) | 2 (2)
platelet count decreased (Blood and lymphatic system disorders) | 7 (9) | 1 (1)
amylase increased (Investigations) | 5 (5) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (3)
fatigue (General disorders) | 11 (14) | 10 (12)
anorexia (Metabolism and nutrition disorders) | 7 (8) | 7 (7)
vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
nausea (Gastrointestinal disorders) | 3 (4) | 1 (1)
lymphocyte count decreased (Investigations) | 2 (2) | 0 (0)
aspartate transaminase increased (Investigations) | 9 (10) | 2 (2)
creatine increased (Investigations) | 3 (4) | 0 (0)
total bilirubin increased (Investigations) | 1 (3) | 0 (0)
pain abdomen (Gastrointestinal disorders) | 2 (3) | 1 (1)
diarrhea (Gastrointestinal disorders) | 4 (7) | 4 (4)
hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
urea nitrogen (Renal and urinary disorders) | 1 (1) | 0 (0)
direct bilirubin increased (Investigations) | 1 (1) | 0 (0)
constipation (Gastrointestinal disorders) | 2 (2) | 5 (5)
thromboembolic event (Vascular disorders) | 2 (2) | 0 (0)
hypothyroidism (Endocrine disorders) | 4 (4) | 4 (4)
decreased T3Free (Investigations) | 2 (2) | 0 (0)
dry mouth (Gastrointestinal disorders) | 2 (2) | 2 (2)
mouth sore (Infections and infestations) | 1 (1) | 0 (0)
Thyroid-stimulating hormone increased (Endocrine disorders) | 2 (2) | 0 (0)
decreased T4 (Investigations) | 1 (1) | 0 (0)
teeth hemorrhage (General disorders) | 1 (1) | 0 (0)
dysgeusia (Nervous system disorders) | 1 (1) | 3 (3)
skin and subcutaneous disease (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
hyperthyroidism (Endocrine disorders) | 2 (2) | 1 (1)
colitis (Gastrointestinal disorders) | 2 (3) | 0 (0)
generalized weakness (General disorders) | 1 (1) | 3 (3)
dry eye (Eye disorders) | 1 (1) | 0 (0)
thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
seizure (Nervous system disorders) | 1 (1) | 0 (0)
hypertension (Cardiac disorders) | 1 (1) | 1 (1)
gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
weight loss (Investigations) | 2 (2) | 2 (2)
hot flashes (Vascular disorders) | 1 (1) | 1 (1)
pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 7 (10)
decreased white blood cells (Investigations) | 1 (1) | 1 (1)
ANC decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
night sweats (Endocrine disorders) | 1 (1) | 0 (0)
tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
thrush (Infections and infestations) | 1 (1) | 0 (0)
hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
chills (General disorders) | 1 (1) | 1 (1)
fever (General disorders) | 0 (0) | 2 (2)
gross hematuria (Renal and urinary disorders) | 0 (0) | 2 (2)
dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
flu like symptoms (General disorders) | 0 (0) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (7)
syncope (Nervous system disorders) | 0 (0) | 1 (1)
nasal congestion (General disorders) | 0 (0) | 1 (2)
dizziness (Nervous system disorders) | 0 (0) | 1 (1)
hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
confusion (Psychiatric disorders) | 0 (0) | 1 (1)
hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
pain throat (General disorders) | 0 (0) | 1 (1)
pain sternum/chest (General disorders) | 0 (0) | 1 (1)
pain bursitis forearm (General disorders) | 0 (0) | 1 (1)
pain face (General disorders) | 0 (0) | 1 (1) — patient fell
neuropathy fingers (Nervous system disorders) | 0 (0) | 1 (1)
memory impairment (Psychiatric disorders) | 0 (0) | 1 (1)
purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
lymph node enlargement (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (2)
myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
blepharitis (Eye disorders) | 0 (0) | 1 (1)
hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
gait disturbance (General disorders) | 0 (0) | 1 (1)
insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
right elbow ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
increased phosphate (Metabolism and nutrition disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-26): https://cdn.clinicaltrials.gov/large-docs/14/NCT02601014/Prot_SAP_000.pdf